CLINICAL TRIAL: NCT01447706
Title: A Phase II Randomized Open Label Study of MM-121 in Combination With Paclitaxel Versus Paclitaxel Alone in Patients With Platinum Resistant/ Refractory Advanced Ovarian Cancers
Brief Title: A Study of MM-121 With Paclitaxel in Platinum Resistant/ Refractory Advanced Ovarian Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merrimack Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MM-121-04-02-08 (ARD11586)
Record Dates: First submitted 2011-10-03; First posted 2011-10-06 (Estimated); Results first posted 2016-05-12 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-04

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: Ovarian Cancer; Platinum-resistant; Platinum-refractory; Fallopian tube cancer; Peritoneal Cancer; Paclitaxel; ErbB3; Phase II; locally advanced/metastatic or recurrent
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Ovarian Neoplasms; Neoplasm Metastasis; Recurrence | interventions — seribantumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paclitaxel (Active Comparator): Standard dosing paclitaxel: 80 mg/m2 QW intravenously)
  Interventions: Drug: Paclitaxel
- MM-121 (SAR256212) + Paclitaxel (Experimental): administered intravenously at 40 mg/kg loading dose on Cycle 1, Week 1 followed by 20 mg/kg QW for all subsequent doses
  Interventions: Drug: MM-121; Drug: Paclitaxel

INTERVENTIONS:
Drug: MM-121 — MM-121 (SAR256212) (IV)
  Other Names: SAR256212
  Arms: MM-121 (SAR256212) + Paclitaxel
Drug: Paclitaxel — Standard dosing Paclitaxel (IV)

SUMMARY:
To determine whether the combination of MM-121 plus paclitaxel is more effective than paclitaxel alone

DETAILED DESCRIPTION:
This is a multicenter, open-label, randomized, Phase II study of MM-121 in patients with platinum resistant or refractory recurrent/advanced ovarian cancers. Up to 210 patients will be randomized (2:1) to receive MM-121 plus paclitaxel or paclitaxel alone.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced/metastatic or recurrent epithelial ovarian cancer, fallopian tube cancer or primary peritoneal cancer
* Received at least one prior platinum based chemotherapy regimen
* Platinum-resistant or refractory
* Eligible for weekly paclitaxel
* Adequate liver and kidney function
* 18 years of age or above

Exclusion Criteria:

* Evidence of any other active malignancy
* History of severe allergic reactions to paclitaxel or other drugs formulated in Cremophor®EL

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2011-10; Primary Completion 2013-09 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor Moyo, MD, Study Director — Merrimack Pharmaceuticals
Locations (10):
- United States (10):
  - Arizona Center for Cancer Care, Glendale, Arizona
  - Pinnacle Oncology, Scottsdale, Arizona
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Wilshire Oncology Medical Group, Corona, California
  - North County Oncology, Oceanside, California
  - Central Coast Medical Oncology, Santa Maria, California
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Carolinas Medical Center/Blumenthal Cancer Center, Charlotte, North Carolina
  - ProMedica Health System, Inc., Toledo, Ohio
  - Chattanooga GYN Oncology, Chattanooga, Tennessee

REFERENCES:
- [Derived] Liu JF, Ray-Coquard I, Selle F, Poveda AM, Cibula D, Hirte H, Hilpert F, Raspagliesi F, Gladieff L, Harter P, Siena S, Del Campo JM, Tabah-Fisch I, Pearlberg J, Moyo V, Riahi K, Nering R, Kubasek W, Adiwijaya B, Czibere A, Naumann RW, Coleman RL, Vergote I, MacBeath G, Pujade-Lauraine E. Randomized Phase II Trial of Seribantumab in Combination With Paclitaxel in Patients With Advanced Platinum-Resistant or -Refractory Ovarian Cancer. J Clin Oncol. 2016 Dec 20;34(36):4345-4353. doi: 10.1200/JCO.2016.67.1891. Epub 2016 Oct 23. PMID 27998236

RESULTS

PARTICIPANT FLOW:
Groups:
- MM-121 + Paclitaxel: MM-121 (20 mg/kg weekly following a 40 mg/kg loading dose) IV infusion over 60 minutes + Paclitaxel (80 mg/m2 weekly) IV infusion over 60 minutes
- Paclitaxel: Paclitaxel: 80 mg/m2 weekly IV infusion over 60 minutes
Period: Overall Study
Arm/Group | MM-121 + Paclitaxel | Paclitaxel
Started | 140 | 83 (3 patients enrolled but not dosed)
Completed | 140 | 80
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MM-121 + Paclitaxel | Paclitaxel | Total
Number analyzed (Participants) | 140 | 83 | 223
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (10.53) | 60.6 (11.85) | 59.6 (11.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 83 | 223
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 5 | 15
  Not Hispanic or Latino | 107 | 62 | 169
  Unknown or Not Reported | 23 | 16 | 39
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian | 111 | 66 | 177
  Black or African American | 2 | 1 | 3
  Alaska Native or American Indian | 0 | 0 | 0
  Asian/Oriental | 1 | 2 | 3
  Native Hawaiian or Pacific Islander | 0 | 0 | 0
  Other | 18 | 8 | 26
  Data Not Reported | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: To determine whether MM-121 + paclitaxel was more effective than paclitaxel alone in prolonging progression-free survival in advanced ovarian cancers resistant or refractory to platinum agents. PFS was a time to event measure, and progression of disease is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), "as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions". Progression free survival was defined as the number of months from the date of randomization to the date of death or progression. If neither death nor progression was observed during the study, PFS data was censored at the last non-progressive disease valid tumor assessment unless the patient was discontinued due to symptomatic deterioration. If this occurred, the patient was counted as having progressive disease (PD).
Time Frame: Time from first dose to date of progression, the longest time frame of 3.9 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MM-121 + Paclitaxel | Paclitaxel
Number analyzed (Participants) | 140 | 80
months | 3.75 [3.48 to 4.63] | 3.68 [2.56 to 5.52]

2. Secondary Outcome: Overall Survival
Description: To determine whether MM-121 + paclitaxel is more effective than paclitaxel alone in prolonging overall survival. This was a time-to-event analysis of time from first dose to date of death.
Time Frame: Time from first dose to date of death, with a median of approximately 13 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MM-121 + Paclitaxel | Paclitaxel
Number analyzed (Participants) | 140 | 83
months | 13.70 [8.77 to NA] — confidence interval upper limit not reached | 10.12 [8.77 to NA] — confidence interval upper limit not reached

3. Post Hoc Outcome: To Explore the Utility of an EGFR Family Receptor-ligand (Heregulin, HRG) as a Predictor of Response to MM-121 and /or Paclitaxel in Formalin Fixed (FFPE) Tumor Samples
Description: Fresh tumor samples were obtained from patients prior to enrollment and formalin-fixed for analysis. Samples were analyzed using RNA-ISH for the expression of the biomarker, heregulin. Progression-free survival was assessed using RECIST v 1.1 to determine whether patients whose tumors express HRG have a lower PFS than those whose tumors do not express HRG, and to assess whether the addition of MM-121 to Paclitaxel can increase PFS in HRG-high patients.
Time Frame: Time from first dose to date of progression, the longest time frame of 3.9 years
Population: Patients with available tissue for RNA-ISH analysis
Measure: Median (95% Confidence Interval); unit: months PFS
Groups:
- HRG High: MM-121 + Paclitaxel; HRG Low: MM-121 + Paclitaxel: MM-121 (20 mg/kg weekly following a 40 mg/kg loading dose) IV infusion over 60 minutes + Paclitaxel (80 mg/m2 weekly) IV infusion over 60 minutes
- HRG High: Paclitaxel; HRG Low: Paclitaxel: Paclitaxel: 80 mg/m2 weekly IV infusion over 60 minutes
Arm/Group | HRG High: MM-121 + Paclitaxel | HRG High: Paclitaxel | HRG Low: Paclitaxel | HRG Low: MM-121 + Paclitaxel
Number analyzed (Participants) | 39 | 19 | 34 | 60
months PFS | 5.7 [3.7 to 7.4] | 3.5 [1.8 to NA] — Confidence interval upper limit not reached | 5.4 [3.6 to NA] — Confidence interval upper limit not reached | 3.5 [2.2 to 3.9]
Statistical Analysis 1: Comparison: HRG High: MM-121 + Paclitaxel vs HRG High: Paclitaxel; Test type: Superiority or Other; p = 0.007, Log Rank; Hazard Ratio (HR) = 0.37, 95% CI 2-sided [0.18 to 0.76]
Statistical Analysis 2: Comparison: HRG Low: Paclitaxel vs HRG Low: MM-121 + Paclitaxel; Test type: Superiority or Other; p = 0.023, Log Rank; Hazard Ratio (HR) = 1.8, 95% CI 2-sided [1.08 to 2.98]

ADVERSE EVENTS:
Time Frame: AEs were collected from a patient's first dose until 30 days after treatment termination. SAEs were collected from time of informed consent until 30 days after termination. If related, events could be reported at any time after termination.
Description: All related AEs ongoing at the time of treatment discontinuation were followed until resolution. Investigators were to report any AEs/SAEs assumed to be related any time, even if occurring more than 30 days after last dose. Though different for each patient, on average, patients could be followed for related AEs/SAEs for ~1 year after termination.
Arm/Group | MM-121 + Paclitaxel | Paclitaxel
Serious Adverse Events (participants affected / at risk) | 59/140 | 25/80
Other Adverse Events (participants affected / at risk) | 140/140 | 79/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MM-121 + Paclitaxel (N=140) | Paclitaxel (N=80)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Adrenal Insufficiency (Endocrine disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 3 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 7 | 4
Small Intestinal Obstruction (Gastrointestinal disorders) | 3 | 3
Subileus (Gastrointestinal disorders) | 3 | 2
Colonic Fistula (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Abdominal Wall Hematoma (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Hemorrhagic ascites (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 2 | 1
Pyrexia (General disorders) | 3 | 4
Disease Progression (General disorders) | 8 | 1
General Physical Health Deterioration (General disorders) | 2 | 1
Infusion Site Extravasion (General disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 0
Device related infection (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Escherichia Sepsis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Abdominal Abscess (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Pelvic Abscess (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Bacteremia (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Post-procedural Fistula (Injury, poisoning and procedural complications) | 1 | 0
Ejection Fraction Decreased (Investigations) | 1 | 0
International Normalized Ratio Increased (Investigations) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Depression (Psychiatric disorders) | 1 | 0
Mental Status Change (Psychiatric disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Renal Pain (Renal and urinary disorders) | 0 | 1
Urinary Fistula (Renal and urinary disorders) | 1 | 0
Female Genital Tract Fistula (Reproductive system and breast disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Toxic Skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Embolism (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1
Pelvic Venous Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MM-121 + Paclitaxel (N=140) | Paclitaxel (N=80)
Diarrhea (Gastrointestinal disorders) | 103 | 34
Fatigue (General disorders) | 63 | 30
Nausea (Gastrointestinal disorders) | 60 | 39
Alopecia (Skin and subcutaneous tissue disorders) | 53 | 26
Vomiting (Gastrointestinal disorders) | 44 | 15
Abdominal pain (Gastrointestinal disorders) | 41 | 20
Anemia (Blood and lymphatic system disorders) | 39 | 24
Decreased appetite (Metabolism and nutrition disorders) | 35 | 20
Asthenia (General disorders) | 34 | 17
Hypokalemia (Metabolism and nutrition disorders) | 34 | 7
Rash (Skin and subcutaneous tissue disorders) | 34 | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 33 | 14
Peripheral Edema (General disorders) | 33 | 16
Hypomagnesemia (Metabolism and nutrition disorders) | 31 | 12
Mucosal Inflammation (General disorders) | 31 | 1
Stomatits (Gastrointestinal disorders) | 31 | 8
Constipation (Gastrointestinal disorders) | 26 | 21
Peripheral neuropathy (Nervous system disorders) | 26 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 25 | 18
Pyrexia (General disorders) | 25 | 21
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 24 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 23 | 7
Dizziness (Nervous system disorders) | 22 | 4
Neutropenia (Blood and lymphatic system disorders) | 22 | 17
Dyspepsia (Gastrointestinal disorders) | 19 | 6
Peripheral Sensory Neuropathy (Nervous system disorders) | 19 | 5
Urinary Tract Infection (Infections and infestations) | 19 | 12
Dysgeusia (Nervous system disorders) | 18 | 16
Erythema (Skin and subcutaneous tissue disorders) | 18 | 2
Headache (Nervous system disorders) | 18 | 13
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 18 | 6
Parasthesia (Nervous system disorders) | 17 | 8
Anxiety (Psychiatric disorders) | 16 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 15 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 15 | 6
Back Pain (Musculoskeletal and connective tissue disorders) | 14 | 12
Dehydration (Metabolism and nutrition disorders) | 14 | 3
Abdominal Distension (Gastrointestinal disorders) | 13 | 8
Abdominal Pain Upper (Gastrointestinal disorders) | 13 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 12
Dry Skin (Skin and subcutaneous tissue disorders) | 13 | 2
Nasopharyngitis (Infections and infestations) | 13 | 7
Pruritis (Skin and subcutaneous tissue disorders) | 13 | 9
Flushing (Vascular disorders) | 12 | 7
Onycholysis (Skin and subcutaneous tissue disorders) | 12 | 4
Hypertension (Vascular disorders) | 11 | 2
Insomnia (Psychiatric disorders) | 11 | 7
Neurotoxicity (Nervous system disorders) | 11 | 5
Rhinitis (Infections and infestations) | 11 | 1
Weight Decreased (Investigations) | 11 | 2
Ascites (Gastrointestinal disorders) | 9 | 7
Depression (Psychiatric disorders) | 9 | 5
Dry Mouth (Gastrointestinal disorders) | 9 | 1
Chills (General disorders) | 8 | 4
Disease Progression (General disorders) | 8 | 1
Hemorrhoids (Gastrointestinal disorders) | 8 | 0
Influenza-like illness (General disorders) | 8 | 3
Intestinal Obstruction (Gastrointestinal disorders) | 8 | 4
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Pain (General disorders) | 8 | 7
Palmer-Plantar Erythrodysasthesia Syndrome (Skin and subcutaneous tissue disorders) | 8 | 0
Vision Blurred (Eye disorders) | 8 | 1
Fall (Injury, poisoning and procedural complications) | 7 | 0
Lacrimation Increased (Eye disorders) | 7 | 2
Leukopenia (Blood and lymphatic system disorders) | 7 | 5
Nail toxicity (Skin and subcutaneous tissue disorders) | 7 | 1
Neutrophil Count Decreased (Blood and lymphatic system disorders) | 7 | 6
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 7 | 9
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 1
Tachycardia (Cardiac disorders) | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less